CLINICAL TRIAL: NCT04946045
Title: The Effect of Sensorimotor Interventions on Feeding Readiness and Oral Feeding Success in Preterm Infants : A Randomized Controlled Study
Brief Title: Feeding Readiness and Oral Feeding Success in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Zühal Çamur, RN, PhD, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Preterm, Feeding Readiness
Record Dates: First submitted 2021-06-23; First posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Preterm; Feeding Behavior; Enteral Feeding Intolerance
Keywords: Preterm; Feeding Readiness; Oral feeding; sensorimotor intervention; neonatal nursing
MeSH Terms: conditions — Premature Birth; Feeding Behavior | interventions — Touch; Palliative Care

STUDY DESIGN:
Intervention Model Description: This research is a randomized controlled study with a control group design with pre-test and post-test measurements from experimental research designs.
Who Masked: Participant, Outcomes Assessor
Masking Description: The "stratified block randomization" method was used to determine which group the preterm infants to be included in the study would be in.
  Stratification was based on gestational age. The phase of inclusion in the study and control groups was carried out by another investigator in order to avoid study bias with block randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention (Tactile/Kinesthetic Stimulation+Nonnutritive Sucking) Group (Experimental): 1. Tactile/Kinesthetic Stimulation (15 min): It was applied 3 times a day, once every 3 hours for 10 days.
  2. Nonnutritive Sucking: It was applied 8 times a day for 10 days with Orogastric (OG) feeding throughout the feeding.
  Interventions: Other: Sensorimotor Interventions (Tactile/Kinesthetic Stimulation+Nonnutritive Sucking)
- Control (Nonnutritive Sucking) Group (No Intervention): 1) Nonnutritive Sucking: Administered during feeding with Orogastric (OG) 8 times a day for 10 days.

INTERVENTIONS:
Other: Sensorimotor Interventions (Tactile/Kinesthetic Stimulation+Nonnutritive Sucking) — Sensorimotor interventions were applied to in preterm infants between 30-33 weeks of age for 10 days. After that, preterms were included in the "Six-phase feeding progression protocol".
  Other Names: Supportive Care
  Arms: İntervention (Tactile/Kinesthetic Stimulation+Nonnutritive Sucking) Group

SUMMARY:
To examine the effects of sensorimotor interventions applied to in preterm infants on readiness for feeding and oral feeding success.

DETAILED DESCRIPTION:
The preterm neonate population cannot potentially be fed orally for a long time in the postnatal period. However, the inability of preterm infants to be fed orally as soon as they are born is not a disease, their adaptation to the external environment of the uterus is more complicated because their physiological functions are not yet mature. This also means long hospital stays for premature babies. Therefore, the American Academy of Pediatrics (AAP) has determined that oral feeding is one of the main criteria for the discharge of the preterm infant from the hospital.

Many studies have been conducted on preterm infants on optimizing oral feeding performance. Studies improve oral feeding skills of preterm infants by applying various sensorimotor interventions and cue-based feeding protocols to improve oral feeding performance. These sensorimotor interventions; non-nutritive sucking (pacifier), sucking-swallowing exercises, oral support, oral stimulation, tactile stimulation, kinesthetic stimulation, sound, smell, audio-visual stimulations, etc. methods were used alone or in combination with these methods.

It has been shown in studies that sensorimotor interventions increase the success of oral feeding in preterms, increase the daily feeding volume, increase weight gain, reduce the cost by shortening the hospital stay, shorten the transition time from gastric feeding to oral/breastfeeding and help mother-infant bonding.

This thesis study was conducted using evidence-based interventions that can facilitate the development of oral feeding skills in preterm infants, the feeding problems they encounter, and their transition from gastric feeding to oral feeding.

ELIGIBILITY:
Inclusion Criteria:

* The mother's milk
* Preterm babies with a gestational age of 30-33 weeks
* No facial deformity,
* No respiratory, cardiovascular, gastrointestinal and neurological disorders or syndromes that would prevent or complicate oral feeding,
* No need for oxygen support,
* There will be preterm infants who are not fed orally, but who are started with tube (Orogastric) feeding.

Exclusion Criteria:

* Transferred to another center during the research,
* Unexpected complication development during the research,
* Occurrence of a pathology that will prevent or complicate oral feeding,
* In cases where there is no voluntary consent of the parent
* The mother is Covid positive

Ages: 30 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Oral Feeding Readiness | 10 days change in T-POFRAS (feeding readiness) after sensorimotor intervention.
  Turkish version of the Preterm Oral Feeding Readiness Assessment Scale (T-POFRAS):It was administered to in preterm infants before and after 10 days of intervention by a neonatal nurse independent of the researcher.

SECONDARY OUTCOMES:
Oral Feeding Success | Change in oral feeding success level according to the 12-day six-phase feeding progression protocol
  Six-phase feeding progression protocol

CONTACTS AND LOCATIONS:
Overall Officials: Zühal Çamur, RN, PhD, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Kınıklı Campus, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No